CLINICAL TRIAL: NCT05617820
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel- Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Estradiol Vaginal Inserts 4 mcg (Teva Pharmaceuticals, Inc.) With IMVEXXY® (Estradiol Vaginal Inserts) (TherapeuticsMD, Inc.) in the Treatment of Dyspareunia in Women With Vulvar and Vaginal Atrophy
Brief Title: Study Comparing Estradiol Vaginal Inserts 4mcg To IMVEXXY ® (Estradiol Vaginal Inerts 4 mcg) In The Treatment Of Dyspareunia in Women With Vulvur and Vaginal Atrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71836003
Record Dates: First submitted 2022-11-07; First posted 2022-11-16 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Dyspareunia
MeSH Terms: conditions — Dyspareunia | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Estradiol vaginal inserts, 4 mcg (Experimental): Estradiol vaginal inserts, 4 mcg. Insert vaginally once daily for 14 days.
  Interventions: Drug: Estradiol
- IMVEXXY® (estradiol vaginal inserts) 4 mcg (Active Comparator): IMVEXXY® (estradiol vaginal inserts) 4 mcg. Insert vaginally once for 14 days.
  Interventions: Drug: Imvexxy
- Placebo vaginal inserts (Placebo Comparator): Placebo vaginal inserts. Insert vaginally once for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol — Vaginal Insert, 4 mcg tablet
  Arms: Estradiol vaginal inserts, 4 mcg
Drug: Imvexxy — Estradiol 4 mcg Vaginal Insert
  Arms: IMVEXXY® (estradiol vaginal inserts) 4 mcg
Drug: Placebo — Vehicle Vaginal Insert
  Arms: Placebo vaginal inserts

SUMMARY:
Randomized, double-blind, placebo-controlled, parallel-designed, multiple-site, bioequivalence study with clinical endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, IRB approved informed consent that meets all criteria of current FDA and local regulations.
2. Females aged 40-75 years inclusive who are postmenopausal, with at least:

   1. 12 months of spontaneous amenorrhea (women <55 year of age with history of hysterectomy without bilateral oophorectomy prior to natural menopause must have Serum follicle-stimulating hormone (FSH) level > 40 mIU/mL); or
   2. 6 months of spontaneous amenorrhea with FSH levels >40mIU/mL; or
   3. At least 6 weeks postsurgical bilateral oophorectomy
3. Have less than or equal to 5% superficial cells on vaginal cytological smear.
4. Vaginal pH > 5.0.
5. Moderate to severe symptom of vaginal pain associated with sexual activity considered the most bothersome vaginal symptom (dyspareunia) of VVA by the patient at screening visit. (i.e., a VVA Symptom Self-Assessment Questionnaire score of 2 or 3) (Appendix B).
6. Women should be sexually active (for example, have sexual activity with vaginal penetration within approximately one month of screening visit).
7. Women should anticipate having sexual activity (with vaginal penetration) during the conduct of the study, and agree to at least one episode of sexual intercourse within study days 10-13.
8. Baseline systolic blood pressure should be no greater than 150 mm Hg and diastolic blood pressure no greater than 90 mm Hg.
9. Normal mammogram completed within 9 months before randomization and a normal clinical breast examination prior to randomization in the study.
10. Patients who have underwent complete Hysterectomy, or in the case of patients with an intact uterus (including patients who underwent a partial hysterectomy) the later must have:

    1. A documented papanicolaou (PAP) smear conducted within 12 months before randomization with no findings that the Investigator believes would contraindicate the use of topical vaginal estradiol.
    2. Documented vaginal ultrasonography results within 3 months before randomization to confirm an inactive endometrial lining, defined as endometrial thickness <4mm.
11. In the opinion of the Investigator, the patient will comply with the protocol and has a high probability of completing the study.

Exclusion Criteria:

1. Premenopasual, perimenopausal, pregnant or lactating patient or planning a pregnancy.
2. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation or could jeopardize the integrity of the study evaluations.
3. Any clinically significant laboratory finding that, in the Investigator's opinion would contraindicate the use of estradiol or compromise patients' safety.
4. Significant history of cholestatic jaundice, hypertension, coronary heart disease or other serious heart problems, uncontrolled diabetes, hypercholesterolemia, hypercalcemia, hypoparathyroidism, hypertriglyceridemia, systemic lupus erythematosus, renal impairment, residual endometriosis posthysterectomy, asthma, epilepsy, migraine, porphyria, hepatic hemangiomas that in the Investigator's opinion would place the study patient at undue risk by participation or could jeopardize the integrity of the study evaluations.
5. History of Protein C, Protein S, or antithrombin deficiency, or other thrombophilic disorder.
6. Patients with known concurrent vaginal infections including but not limited to: Candida albicans, Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhea or Gardnerella vaginalis.
7. Patients with active vaginal herpes simplex infection or have had an outbreak within 40 days before Screening
8. History of sexual abuse that in the opinion of the investigator may interfere with the patient's assessment of vaginal pain with sexual activity.
9. Past or current diagnosis of endometrial hyperplasia.
10. Patients with known, suspected or current history of carcinoma of the breast.
11. Any patients with past or current undiagnosed vaginal bleeding or significant risk factors for endometrial cancer.
12. History of estrogen-dependent neoplasia (e.g., endometrial cancer).
13. Any patients with hypersensitivity to estrogens.
14. Liver impairment or disease or kidney dysfunction or disorder (e.g., chronic renal failure or hepatitis C).
15. History of thrombophlebitis, thrombosis, or thromboembolic disorders.
16. History of cerebrovascular accident, stroke, or transient ischemic attack.
17. History of Myocardial infarction or ischemic heart disease.
18. History or active presence of endocrine disease (except for controlled hypo- or hyper-thyroidism or controlled non-insulin dependent diabetes mellitus). Patients who are on a stable thyroid medication prior to the study should have normal baseline thyroid function test results and expect not to have to change thyroid hormone regimen during the study.
19. Any clinically significant abnormalities on screening physical exam, assessments, ECG, or laboratory tests such as:

    1. Vulvar or vaginal inflammatory condition such as a contact or allergic dermatitis, lichen sclerosis, or other pathological findings.
    2. Presence of suspicious vulvar or vaginal lesions for dysplasia, malignancy, or other pathology other than atrophy.
    3. History of active or chronic pelvic pain.
    4. Painful genital warts or localized areas of ulceration.
    5. Interstitial cystitis.
    6. Unresolved findings suspicious for malignancy on the breast exam; incomplete mammogram result or unresolved findings suggestive of malignant changes or findings requiring follow-up on the pre-study mammogram.
    7. Patients with an intact uterus who have an endometrial thickness of 4mm or greater.
20. Any prescription treatment for vaginal dryness/irritation within 2 weeks before screening or any over the counter or natural remedies, vaginal lubricants or moisturizers within 1 week before screening.
21. Taking inducers of CYP3A4 such as St. John's wort, anticonvulsants, phenylbutazone, rifampin, rifabutin, nevirapine and efavirenz.
22. Taking inhibitors of CYP3A4 such as erythromycin, clarithromycin, ketoconazole, itraconazole, ritonavir, nelfinavir and grapefruit juice.
23. Fasting triglyceride levels > 350 mg/dL.
24. History of radiation therapy or recent (within previous 6 weeks) surgical therapy to the vaginal or cervical areas.
25. Any known or suspected allergies that in the Investigator's opinion would compromise the safety of the patient.
26. Patients who have used vaginal hormonal products (i.e. rings, creams, gels) within the 4 weeks before Screening.
27. Patients who have used transdermal estrogen and/or progestin therapy within the 4 weeks before Screening.
28. Patients who have used oral estrogen, progestin, androgen or selective estrogen receptor modular (SERM) containing drug products within 8 weeks before Screening visit.
29. Intrauterine progestin therapy within 8 weeks before Screening.
30. Use of an intrauterine device within 12 weeks before screening visit.
31. Patients who have used estrogen pellet therapy or progestin implants/ injectable drug therapy within the 6 months before Screening.
32. Patients who have engaged in sexual intercourse or used vaginal douching within 24 hours of the screening visit.
33. Inability to understand the requirements of the study and the relative information or are unable or not willing to comply with the study protocol.
34. Patients who are unable or unwilling to give informed consent.
35. Current history of heavy smoking (more than 15 cigarettes per day) or use of e-cigarettes.
36. Current use of marijuana.
37. Recent history of known alcohol or drug abuse, within one year start of the study.
38. Employees of the Investigator or research center or their immediate family members.
39. Receipt of any drug as part of a research study within 60 days before Screening.
40. Previous participation in this study.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Responder | 15 days
  % Responders where a "Responder" is defined as a patient with: At least a 25% reduction from baseline in the sum of % basal/parabasal + % intermediate cells on vaginal cytology; and Vaginal pH < 5.0 with a change from baseline vaginal pH of at least 0.5
Change in Most Bothersome Symptom | 15 days
  Mean change from baseline to Day 15 in dyspareunia score (the self-identified most bothersome symptom in women with VVA). On a scale of 0 to 3, where 0 = none, 1=mild, 2=moderate and 3 = severe

SECONDARY OUTCOMES:
Treatment Success in Most bothersome symptom | 15 days
  proportion of patients in each treatment group that are considered a Treatment Success at the end of the treatment period evaluated on Day 15. A "Treatment Success" is defined as a score of 0 or 1 on Day 15 for dyspareunia (the self-identified most bothersome symptom at baseline).On a scale of 0 to 3 where 0 = none, 1=mild, 2=moderate and 3 = severe

CONTACTS AND LOCATIONS:
Overall Officials: C Dias, Study Director — Teva Pharmaceuticals USA
Locations (48):
- United States (42):
  - Site 10112, Birmingham, Alabama
  - Site 10146, Chandler, Arizona
  - Site 10103, Sacramento, California
  - Site 10124, Sacramento, California
  - Site 10135, San Diego, California
  - Site 10136, Milford, Connecticut
  - Site 10130, Edgewater, Florida
  - Site 10123, Hialeah, Florida
  - Site 10139, Lake Worth, Florida
  - Site 10115, Leesburg, Florida
  - Site 10138, Maitland, Florida
  - Site 10107, Miami Lakes, Florida
  - Site 10144, Miami Lakes, Florida
  - Site 10101, Miami Springs, Florida
  - Site 10106, New Port Richey, Florida
  - Site 10143, Oldsmar, Florida
  - Site 10129, Ormond Beach, Florida
  - Site 10116, Palm Harbor, Florida
  - Site 10117, Sarasota, Florida
  - Site 10121, Sunrise, Florida
  - Site 10140, Tampa, Florida
  - Site 10119, West Palm Beach, Florida
  - Site 10113, Norcross, Georgia
  - Site 10104, Wichita, Kansas
  - Site 10128, Marrero, Louisiana
  - Site 10109, Metairie, Louisiana
  - Site 10122, New Orleans, Louisiana
  - Site 10105, Saginaw, Michigan
  - Site 10111, Las Vegas, Nevada
  - Site 10147, North Las Vegas, Nevada
  - Site 10126, Lawrenceville, New Jersey
  - Site 10137, New Bern, North Carolina
  - Site 10145, New Bern, North Carolina
  - Site 10134, Philadelphia, Pennsylvania
  - Site 10102, Upper Saint Clair, Pennsylvania
  - Site 10110, North Charleston, South Carolina
  - Site 10118, Chattanooga, Tennessee
  - Site 10142, Beaumont, Texas
  - Site 10120, Fort Worth, Texas
  - Site 10141, Houston, Texas
  - Site 10108, Norfolk, Virginia
  - Site 10154, Seattle, Washington
- El Salvador (2):
  - Site 10148, Santa Tecla, La Libertad Department
  - Site 10149, San Salvador
- Honduras (4):
  - Site 10151, San Pedro Sula
  - Site 10153, San Pedro Sula
  - Site 10150, San Pedro Sula
  - Site 10152, San Pedro Sula